CLINICAL TRIAL: NCT05050162
Title: Randomized Phase II/III Trial of Radiation With Cisplatin at 100 mg/m2 Every Three Weeks Versus Radiation With Weekly Cisplatin at 40 mg/m2 for Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Comparing Cisplatin Every Three Weeks to Cisplatin Weekly When Combined With Radiation for Patients With Advanced Head and Neck Cancer
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: End of Initial Phase of Multi-phase protocol; closed for protocol specified analysis
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-HN009; NCI-2021-08925 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN009 (Other: NRG Oncology); NRG-HN009 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma; Advanced Hypopharyngeal Squamous Cell Carcinoma; Advanced Laryngeal Squamous Cell Carcinoma; Advanced Oropharyngeal Squamous Cell Carcinoma; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (radiation therapy, every 3 week cisplatin) (Active Comparator): Patients undergo radiation therapy over 5 fractions a week for a total of 33-35 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive cisplatin IV once Q3W (on days 1, 22, and 43) during radiation therapy in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, or MRI or PET scan throughout the study.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (radiation therapy, weekly cisplatin) (Experimental): Patients undergo radiation therapy over 5 fractions a week for a total of 33-35 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive weekly cisplatin IV QW for 7 weeks during radiation therapy in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, or MRI or PET scan throughout the study.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Given cisplatin IV every 3 weeks
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: ARM I (radiation therapy, every 3 week cisplatin)
Drug: Cisplatin — Given cisplatin IV weekly
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm II (radiation therapy, weekly cisplatin)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II/III trial compares whether cisplatin given weekly with radiation therapy is better tolerated than cisplatin given every three weeks with radiation therapy for the treatment of head and neck cancer that has spread to other places in the body (advanced). The second part of this study will also help to find out if the cisplatin given weekly approach will extend patients' life by at least the same amount of time as the cisplatin given every three weeks approach. Cisplatin is in a class of medications known as platinum-containing compounds that work by killing, stopping or slowing the growth of cancer cells. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Radiation with low-dose cisplatin given weekly may be effective in shrinking or stabilizing head and neck cancer or preventing its recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether radiation with cisplatin weekly is superior in terms of acute toxicity, as measured by the T-scores (TAME method), to radiation with cisplatin every 3 weeks for patients with locoregionally advanced squamous cell carcinoma of the head and neck (SCCHN). (Phase II) II. To determine whether radiation with cisplatin weekly is non-inferior to radiation with cisplatin every 3 weeks in terms of overall survival (OS) for patients with locoregionally advanced SCCHN. (Phase III) III. To determine whether radiation with cisplatin weekly is superior in terms of acute toxicity, as measured by the T-scores (TAME method), to radiation with cisplatin every 3 weeks for patients with locoregionally advanced SCCHN. (Phase III)

SECONDARY OBJECTIVES:

I. To assess and compare progression-free survival (PFS) between arms. II. To assess and compare locoregional failure and distant metastasis between arms.

III. To assess acute and late toxicity (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).

IV. To assess patient-reported outcomes quality of life (PRO/QOL), as measured by the Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N) (primary PRO), between arms.

V. To assess hearing loss, as measured by audiograms and the modified TUNE grading scale between arms.

VI. To assess hearing loss, as measured by speech audiometry Consonant-Nucleus-Consonant word scores and tympanometry (subject to the modified TUNE grading scale testing results; otherwise, it will be an exploratory objective).

VII. To assess hearing-related QOL as measured by the Hearing Handicap Inventory-Screening (HHIA-S) (secondary PRO), between arms.

VIII. To assess long-term PFS, OS, and toxicity between arms. IX. To assess 3-year restricted-mean survival time for OS and PFS between arms (if long-term update is warranted).

EXPLORATORY OBJECTIVE:

I. To collect blood and tissue specimens for future translational science studies. For instance, to examine how germline and somatic genetic variants, such as TP53, CDKN2A, PIK3CA, PTEN, NFE2L2, and KEAP1, may influence cisplatin-related efficacy and toxicity, and to assess the effect of regular nonsteroidal anti-inflammatory drugs (NSAIDs) use and genomic activation of PIK3CA (mutation or amplification) or loss of PTEN, the negative regulator of PI3K, on disease-free survival or overall survival.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (NON-OROPHARYNGEAL CANCER [OPC]/p16-NEGATIVE OPC group and p16-NEGATIVE OPC/CANCER OF UNKNOWN PRIMARY [CUP] group): Patients undergo radiation therapy over 5 fractions a week for a total of 33-35 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive cisplatin intravenously (IV) once every 3 weeks (Q3W) (on days 1, 22, and 43) during radiation therapy in the absence of disease progression or unacceptable toxicity.

ARM II (NON-OROPHARYNGEAL CANCER [OPC]/p16-NEGATIVE OPC group and p16-NEGATIVE OPC/CANCER OF UNKNOWN PRIMARY [CUP] group): Patients undergo radiation therapy over 5 fractions a week for a total of 33-35 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive cisplatin IV once a week (QW) for 7 weeks during radiation therapy in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT) scan, or magnetic resonance imaging (MRI) or position emission tomography (PET) scan throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of SCCHN of the oropharynx, larynx, hypopharynx, or p16-positive unknown primary prior to registration; specimen from cervical lymph nodes with a well-defined primary site documented clinically or radiologically is acceptable; in patients with carcinoma of unknown primary this will be sufficient for pathologic confirmation without a clinically or radiographically defined primary site

  * For patients with oropharyngeal cancer (OPC)/cancer of unknown primary (CUP):

P16 status based on local site immunohistochemical tissue staining is required. A cell block obtained from a fine needle aspiration (FNA) biopsy specimen may be used as the sole diagnostic tissue. Centers are encouraged to contact the pathology chair for clarification.

* Note: Institutions must screen patients for p16 status by immunohistochemistry (IHC) in order to be eligible for the trial using a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. A rigorous laboratory accreditation process similar to the United States (U.S.) CLIA certification, such as the provincial accreditation status offered by the Ontario Laboratory Accreditation (OLA) Program in Canada, the College of American Pathologists (CAP), or an equivalent accreditation in other countries, is acceptable.

  * The p16 results must be reported on the pathology report being submitted. The p16 positivity is defined as > 70% of tumor cells showing strong nuclear and/or cytoplasmic immunostaining with p16 antibody.
  * For patients with laryngeal and hypopharyngeal primaries: Analysis of p16 status is NOT required.

    * Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations. Simple tonsillectomy or local excision of the primary without removal of nodal disease is permitted, as is excision removing gross nodal disease but with intact primary site. Limited neck dissections retrieving =< 4 nodes are permitted and considered as non-therapeutic nodal excisions
    * Clinical stage (American Joint Committee on Cancer [AJCC], 8th ed.), including no distant metastases based on the following diagnostic workup:
  * History/physical examination within 60 days prior to registration
  * One of the following imaging studies is required within 60 days prior to registration:
* Computed tomography (CT) scan of neck (diagnostic quality with contrast, unless contraindicated) OR
* Magnetic resonance imaging (MRI) of the neck (diagnostic quality with contrast, unless contraindicated) OR
* Fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/CT of the neck; the CT component must be of diagnostic quality with contrast, unless contraindicated.

  * Note: A diagnostic quality CT or MRI with contrast or FDG-PET/CT scan of neck performed for the purposes of radiation planning may serve as both staging and planning tools

    * One of the following imaging studies is required within 60 days prior to registration:
* FDG-PET/CT of the chest; FDG-PET/CT scan is strongly preferred and highly recommended to be used for eligibility OR
* Chest CT

  * Exam with laryngopharyngoscopy (mirror or in office direct procedure acceptable) within 70 days prior to registration;
* Eligibility by patient cohort;

  * Non-OPC/p16-negative OPC Cohort; Tumor Site: Larynx/Hypopharynx; Clinical Staging (AJCC, 8th ed.): T3-4 N0 or T1-4 N1-3 T2 N0 (hypopharynx only)
  * Tumor Site: p16-negative OPC; Clinical Staging (AJCC, 8th ed.): T2N1, T1-4 N2-3, or T3-4 N0-1
* p16-positive OPC/CUP Cohort;

  * Tumor Site: OPC; Smoking Status: =< 10 pack-years; Clinical Staging (AJCC, 8th ed.): T1-3 N2-3 or T4 N0-3
  * Tumor Site: OPC; Smoking Status: > 10 pack-years; Clinical Staging (AJCC, 8th ed.): T1N2-3, T2N1-3, or T3-4 N0-3
  * Tumor Site: CUP; Smoking Status: Any; Clinical Staging (AJCC, 8th ed.): T0 N2-3 Note: Cigar and pipe tobacco consumption is not included in calculating the lifetime pack-years. Marijuana consumption is likewise not considered in this calculation. There is also no clear scientific evidence regarding the role of chewing tobacco-containing products in oropharyngeal cancer, although this is possibly more concerning given the proximity of the oral cavity and oropharynx. In any case, investigators should not count use of non-cigarette tobacco products in the pack-years calculation.

    * Age >= 18
    * Zubrod (Eastern Cooperative Oncology Group [ECOG]) performance status of 0-1 within 14 days prior to registration
    * Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 30 days prior to registration)
    * Platelets >= 75,000 cells/mm^3 (within 30 days prior to registration)
    * Hemoglobin >= 8.0 g/dL (within 30 days prior to registration)

      * Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dL is acceptable)
    * Calculated creatinine clearance (CrCl) >= 50 mL/min by the Cockcroft-Gault formula (within 30 days prior to registration)
    * Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 30 days prior to registration) (not applicable to patients with known Gilbert's syndrome)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x institutional ULN (within 30 days prior to registration)
    * Known human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and CD4 T Cell count > 200 cells/mm^3 are eligible for this trial. Testing is not required for entry into protocol
    * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
    * Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
    * Willing to use highly effective contraceptives for participants of childbearing potential (participants who may become pregnant or who may impregnate a partner) during therapy and for 14 months (females); for 11 months (males) following last dose of cisplatin; this inclusion is necessary because the treatment in this study may be significantly teratogenic.
    * The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients with oral cavity cancer, nasopharynx cancer, or p16-negative cancer of unknown primary (CUP)
* Recurrence of the study cancer
* Definitive clinical or radiologic evidence of distant metastatic disease
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable, however, any prior exposure to cisplatin is excluded
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity defined as follows:

  * Unstable angina requiring hospitalization in the last 6 months
  * Myocardial infarction within the last 6 months
  * New York Heart Association Functional Classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  * Persistent grade 3-4 (CTCAE version 5.0) electrolyte abnormalities that cannot be reversed despite replacement as indicated by repeat testing
  * Patient must not have an active infection requiring IV antibiotics prior to registration;
  * Other chronic renal disease like nephrotic syndrome, that could be worsened by cisplatin therapy
  * History of allogenic organ transplantation
  * Any symptomatic peripheral sensory neuropathy grade >= 2 (CTCAE version 5.0);
* Pregnancy and individuals unwilling to discontinue nursing
* History of hypersensitivity to cisplatin or platinum-containing compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1714 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute toxicity (Phase II) | Up to 180 days post-treatment
  Measured by the T-scores.
Overall survival (OS) (Phase III) | From randomization to death of any cause, assessed up to 9 years
  OS rates will be estimated using the Kaplan-Meier method.
Incidence of acute toxicity (Phase III) | Up to 180 days post-treatment
  Measured by the T-scores.

SECONDARY OUTCOMES:
Locoregional failure rates | Up to 9 years
Distant metastasis | Up to 9 years
Progression-free survival (PFS) | From randomization to locoregional failure, distant metastasis, or death due to any cause, whichever occurs first, assessed up to 9 years
  PFS rates will be estimated using the Kaplan-Meier method and between-arm differences compared using the log-rank test with a two-sided alpha of 0.05 (Kaplan 1958).
Restricted mean survival time (RMST) for OS | At 3 years
  Compared using a Wald-type test based on Kaplan-Meier estimates. Adjusted RMST estimates at 3 years and 95% confidence intervals will be provided using RMST regression with pseudo-observations.
RMST for PFS | At 3 years
  Compared using a Wald-type test based on Kaplan-Meier estimates. Adjusted RMST estimates at 3 years and 95% confidence intervals will be provided using RMST regression with pseudo-observations.
Incidence of acute toxicity | Up to 180 days post-treatment
  Measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of late toxicity | Up to 9 years
  Measured by CTCAE v5.0.
Incidence of late toxicity | Up to 9 years
  Measured by the A-scores.
Quality of life | At 6 months post-radiation therapy
  Measured by Functional Assessment of Cancer Therapy Head and Neck.
Hearing loss | At 6 months post-radiation therapy
  Measured by Hearing Handicap Inventory for Adults-Screening.
Hearing loss (cochleotoxicity) | At 6 months post-radiation therapy
  Measured by audiograms and the modified TUNE grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Harari, Principal Investigator — NRG Oncology
Locations (370):
- United States (361):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - AdventHealth Parker, Parker, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - FHCC Overlake, Bellevue, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (5):
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Ireland (2):
  - Saint Lukes Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
- Kantonsspital Aarau, Aarau, Switzerland